CLINICAL TRIAL: NCT05237453
Title: Pulmonary Magnetic Resonance-guided Online Adaptive Radiotherapy of Locally Advanced Non-Small Cell Lung Cancer
Acronym: PUMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: University Hospital Tuebingen (Other); Ludwig-Maximilians - University of Munich (Other); German Cancer Research Center (Other)
Responsible Party: Principal Investigator, Juergen Debus, Head of Department, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RadOnk-PUMA_2021
Record Dates: First submitted 2022-01-13; First posted 2022-02-14 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: lung cancer; adaptive Radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR-guided adaptive radiotherapy (Experimental): Patients receive Photon radiotheray as an MR-guided adaptive radiotherapy
  Interventions: Radiation: Photons

INTERVENTIONS:
Radiation: Photons — MR-guided adaptive radiotherapy

SUMMARY:
MR-guided radiotherapy is an innovative technique which supports sophisticated approaches towards pulmonary adaptive radiotherapy (ART). Such individualized treatment approaches can lead to reduced toxicity and potentially better local tumor control for patients with LA-NSCLC in the future. PUMA is an early clinical trial, which aims to demonstrate the feasibility of MR-guided online ART to locally-advanced NSCLC. In a second step, the investigators aim to use the data from this feasibility trial to design and launch a further phase I/II clinical study that directly compares the benefits of MR-guided online ART of LA-NSCLC to CT-based (A)RT approaches.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) is very common and carries the highest mortality of all malignant diseases (350.000 - 400.000 deaths per year in the European Union). In specific, the 5-year overall survival rate of locally-advanced NSCLC (LA-NSCLC) is merely 20%. One reason for this dismal prognosis is the lack of effective treatment options. Since most patients with LA-NSCLC are not candidates for a tumor resection, definitive (chemo)radiotherapy (C)RT with consecutive immunotherapy (IT) is the treatment of choice according to national and international guidelines. However, local tumor relapse remains a major pattern of recurrence in approx. 30% of cases. Furthermore, many patients cannot benefit from chemotherapy due to multiple comorbidities, and application of IT requires an initial tumor response to (C)RT and absence of higher-grade pulmonary toxicity. Consequently, radiotherapy is a cornerstone in the locally ablative treatment of LA-NSCLC and essentially influences the course of the further treatment. MR-guided radiotherapy is an innovative technique which supports sophisticated approaches towards pulmonary adaptive radiotherapy (ART). Such adaptive radiation approaches allow highly individualized thoracic radiotherapy with dose distributions tailored to the interfractional changes in tumor geometry and anatomy of surrounding OARs. Therefore, MR-guided ART has the potential to optimize the balance between intensified target volume dose and sparing of vulnerable OARs. This prospective, multicenter clinical trial is desinged to demonstrate the clinical feasibility and gain first data on the safety of MR-guided online ART to LA-NSCLC. Based on the investigators extensive experience with MR-guided RT of early-stage NSCLC and lung metastases, the invesitgators hypothesize that MR-guided online ART to LA-NSCLC can be performed successfully in ≥ 80% of patients with a mean time < 90 minutes. The investigators plan to include 30 patients with LA-NSCLC in Union for International Cancer Control (UICC) stage IIIA-C at three German university hospitals (Uniklinikum Heidelberg, Uniklinikum LMU München, Uniklinikum Tübingen). Patients will receive MR-guided online ART, which includes gated dose delivery as well as online plan adaptation once weekly or in case major anatomical changes are detected on daily MR-imaging. Patients will be followed-up to assess toxicity, tumor control (by means of thoracic CT- and MR-imaging) and patient-reported outcomes for 24 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven non-small cell lung cancer (NSCLC)
* Stage III A - C according to the 8th edition of the Union for International Cancer Control (UICC) TNM classification
* Indication for definitive thoracic chemoradiotherapy
* Age ≥ 18 years
* ECOG 0 - 2
* Adequate pulmonary function for chemoradiotherapy confirmed by a current pulmonary function test (≤ 6 weeks from treatment start)
* Ability to lie still on the MR-linac table for at least one hour
* Ability to hold one's breath for at least 20 seconds
* Successful completion of an MR-guided treatment simulation
* For women with childbearing potential: adequate contraception
* Ability of the patient to understand character and individual consequences of the clinical trial
* Written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

* Involvement of supraclavicular lymph nodes (supraclavicular N3)
* Additional pulmonary lesions (T3 - 4 due to additional lesion in the same or another lobe)
* Previous radiotherapy of the lung and mediastinum, if previous and current target volumes overlap
* Patients who have not yet recovered from acute toxicities of prior therapies
* Contraindications against performing MRI scans (e.g. pacemakers or other implants making MRI impossible)
* Pregnant or lactating women
* Participation in another competing clinical study or observation period of competing trials
* Refusal of the patients to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
clinical feasibility -1- | through study completion, an average of 2 years
  successfully completed online adapted RT fractions
clinical feasibility -2- | through study completion, an average of 2 years
  treatment time for online adapted RT fractions

SECONDARY OUTCOMES:
acute side effects | 3 months from treatment start
  changes in toxicity according to CTCAE V5.0
subacute side effect | 6 months from treatment start
  changes in toxicity according to CTCAE V5.0
chronic side effect | through study completion, at least 24 months
  changes in toxicity according to CTCAE V5.0
Local tumor control | through study completion, at least 24 months
  time from treatment start until in-field tumor recurrence
Progession free survival | through study completion, at least 24 months
  time from treatment start until death or progression of tumor disease
Overall survival | through study completion, at least 24 months
  time from treatment start until death
Longitudinal pulmonary function | through study completion, at least 24 months
  changes in forced exspiratory volume in 1st second (FEV1s), vital capacity (vc), etc.

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Debus, Prof, Principal Investigator — University Hospital Heidelberg
Locations (3):
- Germany (3):
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Ludwig-Maximilian-Universität München, Münich, Bavaria
  - University Hospital of Heidelberg, Radiation Oncology, Heidelberg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Regnery S, de Colle C, Eze C, Corradini S, Thieke C, Sedlaczek O, Schlemmer HP, Dinkel J, Seith F, Kopp-Schneider A, Gillmann C, Renkamp CK, Landry G, Thorwarth D, Zips D, Belka C, Jakel O, Debus J, Horner-Rieber J. Pulmonary magnetic resonance-guided online adaptive radiotherapy of locally advanced: the PUMA trial. Radiat Oncol. 2023 May 4;18(1):74. doi: 10.1186/s13014-023-02258-9. PMID 37143154